CLINICAL TRIAL: NCT00224796
Title: A Randomized, Controlled Multicenter Trial of Vacuum Assisted Closure® Therapy in the Treatment and Blinded Evaluation of Amputation Wounds of the Diabetic Foot
Brief Title: Trial of Vacuum Assisted Closure® Therapy in Amputation Wounds of the Diabetic Foot
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAC2001-07
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot
Keywords: Wound closure; Foot salvage; Accelerated healing; Amputation Wounds of the Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

INTERVENTIONS:
Device: V.A.C. ® System

SUMMARY:
The purpose of this study is to compare the effectiveness of Vacuum Assisted Closure® (V.A.C.®) Therapy to moist wound therapy of amputation wounds of the diabetic foot. The primary objective is to determine the effect of V.A.C.® Therapy on the incidence of complete wound closure. Secondary objectives include evaluating the acceleration of wound closure, facilitation of surgical closure, incidence of foot salvage, and incidence of wound complications.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a diabetic foot amputation wound up to the transmetatarsal region of the foot
2. Evidence of adequate perfusion by one of the following on the affected extremity, (within the past 60 days):

   * Dorsum transcutaneous oxygen test (TcPO2) with results of ≥30 mmHg, or
   * Ankle brachial index (ABIs) with results of ≥0.7 and ≤1.2 and toe pressures with results of ≥30 mmHg, or
   * Doppler arterial waveforms, which are triphasic or biphasic at the ankle in the affected leg.
3. Age ≥ 18 years of age
4. HbA1c ≤ 12% (collected within the last 90 days.)
5. Evidence of adequate nutrition by one of the following:

   * Lab results reflecting Pre-Albumin ≥16 mg/dl and Albumin level is ≥3 g/dl (during the seven days prior to the study period), or
   * A nutritional consult will be done and with appropriate supplementation started. Proper documentation on (case report forms)CRFs is needed.

Exclusion Criteria:

1. Patients with recognized active Charcot abnormalities of the foot, as evidence by clinical symptoms that interfere with either randomized treatment group
2. Wounds resulting from electrical, chemical, or radiation burns, or venous insufficiency
3. Untreated infection or cellulitis at site of target wound
4. Presence of untreated osteomyelitis
5. Collagen vascular disease
6. Malignancy in the wound
7. Presence of necrotic tissue in the wound
8. Uncontrolled hyperglycemia
9. Concomitant medications that include (washout period of 30 days for corticosteroids, immunosuppressive medications, or chemotherapy)
10. Prior V.A.C.® therapy within 30 days.
11. Current or prior normothermic (Warm-UP®) or hyperbaric oxygen (HBO) therapy within 30 days.
12. Current or prior treatment with recombinant or autologous growth factor products within the past 30 days. (Examples: Regranex or Procuren)
13. Current or prior treatment with skin or dermal substitutes and dressings (Examples: Apligraf, Dermagraft, or Integra) with living cells capable of producing growth factors (Example: Oasis) within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146
Dates: Start 2002-05; Study Completion 2005-10

PRIMARY OUTCOMES:
To determine the effect of V.A.C. ® Therapy on the incidence of complete wound closure.

SECONDARY OUTCOMES:
To determine the effect of V.A.C. ® Therapy on the accelerated wound closure or facilitation of surgical closure
To determine the incidence of foot salvage, as defined by retention of transmetatarsal amputation with no further revisions at end of study
To determine the change in wound area over time
To determine the incidence of complications
To determine the effect of V.A.C. ® Therapy on the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, DPM, Principal Investigator — Rosalind Franklin University

REFERENCES:
- [Background] Holzer SE, Camerota A, Martens L, Cuerdon T, Crystal-Peters J, Zagari M. Costs and duration of care for lower extremity ulcers in patients with diabetes. Clin Ther. 1998 Jan-Feb;20(1):169-81. doi: 10.1016/s0149-2918(98)80044-1. PMID 9522113
- [Background] Glover JL, Weingarten MS, Buchbinder DS, Poucher RL, Deitrick GA 3rd, Fylling CP. A 4-year outcome-based retrospective study of wound healing and limb salvage in patients with chronic wounds. Adv Wound Care. 1997 Jan-Feb;10(1):33-8. PMID 9204802
- [Background] Bild DE, Selby JV, Sinnock P, Browner WS, Braveman P, Showstack JA. Lower-extremity amputation in people with diabetes. Epidemiology and prevention. Diabetes Care. 1989 Jan;12(1):24-31. doi: 10.2337/diacare.12.1.24. PMID 2714164
- [Background] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970
- [Background] Banwell PE. Topical negative pressure therapy in wound care. J Wound Care. 1999 Feb;8(2):79-84. doi: 10.12968/jowc.1999.8.2.25844. No abstract available. PMID 10232203
- [Background] Mullner T, Mrkonjic L, Kwasny O, Vecsei V. The use of negative pressure to promote the healing of tissue defects: a clinical trial using the vacuum sealing technique. Br J Plast Surg. 1997 Apr;50(3):194-9. doi: 10.1016/s0007-1226(97)91369-2. PMID 9176007
- [Background] Sibbald RG. Venous leg ulcers. Ostomy Wound Manage. 1998 Sep;44(9):52-64; quiz 65-6. PMID 9866605
- [Result] Armstrong DG, Lavery LA; Diabetic Foot Study Consortium. Negative pressure wound therapy after partial diabetic foot amputation: a multicentre, randomised controlled trial. Lancet. 2005 Nov 12;366(9498):1704-10. doi: 10.1016/S0140-6736(05)67695-7. PMID 16291063
- [Derived] Armstrong DG, Lavery LA, Boulton AJ. Negative pressure wound therapy via vacuum-assisted closure following partial foot amputation: what is the role of wound chronicity? Int Wound J. 2007 Mar;4(1):79-86. doi: 10.1111/j.1742-481X.2006.00270.x. PMID 17425550